CLINICAL TRIAL: NCT04456452
Title: A Randomized Controlled Trial to Evaluate the Safety of Intravenous Ampion™ in Adult COVID-19 Patients Requiring Oxygen Supplementation
Brief Title: Study of Ampion for the Treatment of Adult COVID-19 Patients Requiring Oxygen Supplementation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP-016
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — aspartyl-alanyl-diketopiperazine; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ampion (Experimental): Ampion
  Interventions: Biological: Ampion; Other: Standard of Care
- Standard of Care (Other): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Ampion — Ampion, administered by intravenous infusion
  Arms: Ampion
Other: Standard of Care — Standard of Care

SUMMARY:
This is a Phase 1 randomized study to evaluate the safety, tolerability and efficacy of IV Ampion in improving the clinical course and outcomes of patients hospitalized with COVID-19 infection who require supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years to 89 years old (inclusive).
2. Hospitalized and diagnosed with COVID-19, as evaluated by PCR test confirming infection with SARS-COV-2.
3. Patient is receiving supplemental oxygen (e.g. oxygen saturation (SpO2) <88%, labored breathing, increased respiratory rate, dyspnea on rest or exertion).
4. A signed informed consent form from the patient or the patient's legal representative must be available.

Exclusion Criteria:

1. In the opinion of the clinical team, progression to death is imminent and inevitable, irrespective of the provision of treatments.
2. Patient has severe chronic obstructive pulmonary disease (COPD), chronic renal failure, or significant liver abnormality (e.g. cirrhosis, transplant, etc.).
3. Patient is on chronic immunosuppressive medication.
4. As a result of the medical review and screening investigation, the Principal Investigator considers the patient unfit for the study.
5. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion) or excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
6. Patient has known pregnancy or is currently breastfeeding.
7. Participation in another clinical trial.
8. Baseline QT prolongation.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Primary endpoint at day 5
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Colorado Springs, Colorado, United States